CLINICAL TRIAL: NCT03388710
Title: Consultant Anesthesiology
Brief Title: Position of the Endotracheal Tube Cuff in Relation to Cricoid in Children.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Tariq Wani, Consultant Anesthesiology, King Fahad Medical City
Other Study IDs: KFMC
Record Dates: First submitted 2017-12-25; First posted 2018-01-03 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: D009863
Keywords: airway, children, endotracheal tube, cuff
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: XRay — Xray to confirm the location of the endotracheal tube

SUMMARY:
To verify the exact location of cuff of the endotracheal tube in children.

DETAILED DESCRIPTION:
The exact location of the cuff of the endotracheal tube in children has not been studied. This study is the first attempt to verify the position of the cuff in the airway with relation to cricoid.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 8 years

Exclusion Criteria:

* Any airway pathology

Ages: 1 Month to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children for any surgical procedure requiring endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Cuff position | 6 months
  Location of the cuff of the ETT

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Wani, MD, Principal Investigator — Consultant
Locations (1):
- King Fahad Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided